CLINICAL TRIAL: NCT01711944
Title: Online Implementation of Problem Solving Skills Training for Mothers of Newly Diagnosed Childhood Cancer Patients
Brief Title: Online Problem Solving Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: M.D. Anderson Cancer Center (Other); University of Texas, El Paso (Other); University of Colorado, Denver (Other); University of Pittsburgh (Other); Rutgers Cancer Institute of New Jersey (Other); Children's Hospital Los Angeles (Other); St. Jude Children's Research Hospital (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, OJ Sahler, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01CA159013-01A1 (NIH); R01CA159013-01A1 (NIH)
Record Dates: First submitted 2012-09-29; First posted 2012-10-22 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Childhood Cancer
Keywords: childhood cancer; Internet communication; parents; caregivers; problem solving
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online PSST (Experimental): An online version of Problem-Solving Skills Training (PSST) will be compared to standard (face-to-face) PSST
  Interventions: Behavioral: Problem-Solving Skills Training
- Face-to-Face PSST (Active Comparator): This is an 8-session face-to-face Problem-Solving Skills Training intervention
  Interventions: Behavioral: Problem-Solving Skills Training

INTERVENTIONS:
Behavioral: Problem-Solving Skills Training — 8-session manualized intervention to provide problem-solving skills training in the context of childhood cancer.
  Other Names: PSST; Bright IDEAS; Online PSST; Standard or face-to-face PSST

SUMMARY:
Parents of children newly diagnosed with cancer experience depression and anxiety, especially in the first several months of treatment. Bright IDEAS, an 8-session problem-solving skills training (PSST) program has been used in studies with more than 900 mothers including more than 125 monolingual Spanish-speaking mothers. It has been shown to significantly decrease mothers' distress and to particularly benefit Latina immigrants. This past spring, the NCI/NIH designated Bright IDEAS as a Research-Tested Intervention Program and has included it in the National Registry of Evidence-based Programs and Practices. To date, Bright IDEAS has been available to mothers at only a few cancer centers with specially trained personnel. This proposal is designed to bring Bright IDEAS on-line to make it available to mothers and fathers 24/7 anywhere with Internet access. The investigators will carefully analyze acceptability and use to gain insight into the most promising ways of disseminating interventions like Bright IDEAS using Internet, Internet II, and other emerging technologies.

DETAILED DESCRIPTION:
Research and experience document that caregivers of children with cancer encounter extraordinary stresses during the child's illness. These stresses are particularly severe during diagnosis and early therapy and can interfere significantly with a caregiver's ability to make reasoned and timely decisions on their child's behalf. With increasing survivor rates, it has become evident that decisions made in the early stages of cancer management can have profound long-term effects, adding to the distress caregivers feel trying to make the "right" decisions. Too help mothers of newly diagnosed children cope more effectively with these challenges, the investigators conducted randomized controlled trials (R25CA65520, R01CA098954) to develop, field test, and evaluate the efficacy of the Bright IDEAS paradigm of problem-solving skills training (PSST), a cognitive-behavioral therapy shown to decrease anxiety and depression - two symptoms of post-traumatic stress commonly experienced among this group of mothers. Our findings clearly show that PSST significantly increases problem-solving skills (primary effect) and decreases negative affectivity (secondary effect) in mothers from a variety of racial, ethnic, and socioeconomic backgrounds. Particularly powerful and long-lasting effects were noted in Spanish-speaking mothers, an especially underserved population. In March 2010, the NCI designated Bright IDEAS as a Research-based Therapy/Intervention Program (RTIP) and entered it into the National Registry of Evidence-based Programs and Practices (NREPP). As an 8-session, in-person intervention, Bright IDEAS is labor intensive and, to date, has only been available at a few institutions with trained personnel. However, as a part of the RTIPs evaluation process, the Dissemination Capability of Bright IDEAS was rated 5/5. This proposal is designed to meet the challenge inherent in this perfect score. The investigators will also immediately broaden the scope of users by including fathers as eligible participants in this study of a new delivery paradigm the investigators believe they will find appealing. Aim 1 is implementation of an engaging, easy-to-use on-line version of Bright IDEAS that would be available 24/7 to any person anywhere who has access to the Internet. Aim 2 is the use of "Diffusion of Innovations" theory to craft a framework for disseminating not only Bright IDEAS but other similar interventions with the greatest effectiveness and efficiency. In past studies, the investigators have shown that the human element (time and attention) inherent in in-person interventions is effective in bringing immediate relief of distress but not sufficient to maintain its benefits over time. In contrast, mothers receiving PSST increase their skills and continue to improve their sense of well-being 3 months after the intervention. What the investigators have not investigated is whether a computer-based intervention is as effective as (not inferior to) an in-person intervention. The results will have significant implications for future dissemination strategies, especially the use of Internet II and other emerging technologies.

ELIGIBILITY:
Inclusion Criteria: Subjects will be drawn from the pool of all parents who are primary caregivers of children diagnosed with any form of cancer 4-16 weeks prior to contact about the Problem Solving Skills Training intervention and cared for at one of the 4 data collection sites. No attempt will be made to stratify the sample by any particular demographic variables (e.g., age, ethnic background, or type of cancer diagnosed in their child), except that monolingual Spanish-speaking parents will be specifically recruited to provide adequate representation for statistical analysis at Childrens Hospital Los Angeles and UT/MD Anderson Cancer Center. Goal: 20% total enrollment.

Exclusion Criteria: Parents of children with cancer will be excluded if (1) they do not read or speak English or Spanish; (2) their child is in severe a medical crisis, as determined by the oncologist, or (3) they live a prohibitive distance to complete the intervention (typically, >50 miles from the Center) and do not have access to a telephone for phone intervention sessions. Internet access will be facilitated as part of the e-PSST intervention arm. These exclusionary criteria are identical to our previous work; <10% of eligible mothers have been excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2012-07; Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Social Problem Solving Skills Inventory | Baseline (T1), post intervention (3 months; T2), 3 months post intervention (6 months; T3)
  This is a well validated assessment of problem-solving strategies and positive or negative orientation to problem solving.

SECONDARY OUTCOMES:
Profile of Mood States | Baseline (T1); post intervention (3 months; T2); 3 months post intervention (6 months; T3)
  This is a well validated measure of depression and anxiety
Patient Health Questionnaire (PHQ9) | Baseline (T1), post intervention (3 months; T2), 3 months post intervention (6 months; T3)
  A 9-item self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ9 is the depression module which rates each of the nine DSM-IV criteria as 0 (not at all) to 3 (nearly every day). It will be used in place of the Beck Depression Inventory.

OTHER OUTCOMES:
Impact of Event Scale-Revised | Baseline (T1); post intervention (3 months; T2); 3 months post intervention (6 months; T3)
  This is a well-validated assessment of the impact of a specified event (in this case, the diagnosis of cancer in a child)
Bidimensional Acculturation Scale for Hispanics | Baseline (T1); post intervention (3 months; T2); 3 months post intervention (6 months; T3)
  This is a well-validated measure of the degree to which an individual born in another country has adopted the customs of their new country
Hispanic Stress Inventory | Baseline (T1); post intervention (3 months; T2); 3 months post intervention (6 months; T3)
  This is a well validated assessment of the social, financial, and emotional ramifications associated with being a minority individual (in this case, Hispanic).
Current Problems Inventory | Baseline (T1), post intervention (3 months; T2), 3 months post intervention (6 months; T3)
  The Current Problems Inventory was developed by the investigators to provide examples of the kinds of problems commonly encountered in families with a child with cancer. This form has been completed by participants at T1 in all studies of Bright IDEAS PSST to date. During this project, the CPI will be given at T1, T2, and T3 to monitor change over time.
Demographic Information | Baseline (T1)
  Includes information about the child with cancer (age, diagnosis, date of diagnosis), parental age, marital status, educational level, occupational prestige of the family, and previous experience with the Internet.
Impact of Event Scale-Revised (IES-R) | Baseline (T1), post intervention (3 months; T2), 3 months post intervention (6 months; T3)
  A 22-item self-report measuring perceived post-traumatic stress, includes three subscales (intrusion, avoidance, and hyperarousal) that assess PTS symptoms (PTSSx) during the past week experienced in response to a specific event. Widely used to measure PTSSx associated with events such as diagnosis with cancer. Internal consistency reliabilities of the intrusion, avoidance, and hyperarousal subscales are .91, .84, and .90, respectively.
Credibility/Expectancy | After the first face-to-face PSST or ePSST session and after the fourth face-to-face PSST session or four weeks after the first ePSST session
  Credibility is measured along four dimensions and expectancy is rated on a scale of 0 to 100. These rating scales were developed by the investigators specifically for this purpose and used in our most recent previous study.
User Satisfaction | Post intervention (3 months; T2)
  Will be assessed using a 21-item questionnaire developed by the investigators to address intervention-specific and website-specific issues. Only the first five questions and the open-ended questions modified for the face-to-face group (specific to Bright IDEAS itself) will be completed by participants receiving the standard intervention. The questionnaire will be administered at T2.

CONTACTS AND LOCATIONS:
Overall Officials: Olle Jane Z Sahler, MD, Principal Investigator — University of Rochester
Locations (6):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Rochester Medical Center, Rochester, New York
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Texas/MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Phipps S, Fairclough DL, Noll RB, Devine KA, Dolgin MJ, Schepers SA, Askins MA, Schneider NM, Ingman K, Voll M, Katz ER, McLaughlin J, Sahler OJZ. In-person vs. web-based administration of a problem-solving skills intervention for parents of children with cancer: Report of a randomized noninferiority trial. EClinicalMedicine. 2020 Jun 27;24:100428. doi: 10.1016/j.eclinm.2020.100428. eCollection 2020 Jul. PMID 32637901